CLINICAL TRIAL: NCT04183686
Title: Single-center, Double-blind, Randomized, Placebo-controlled Phase 1 Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Single- and Multiple-ascending Doses of ACT-1014-6470 in Healthy Subjects, Including Food Effect, Mass Balance, and Metabolite Profiling
Brief Title: A Study to Examine the Safety, Tolerability, and Pharmacokinetics of Single- and Multiple-ascending Doses of ACT-1014-6470 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: ID-087-101
Record Dates: First submitted 2019-11-26; First posted 2019-12-03 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Healthy
MeSH Terms: interventions — ACT-1014-6470; Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide

STUDY DESIGN:
Intervention Model Description: Single-center, double-blind, randomized, placebo-controlled Phase 1 study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Part A (SAD): Dose A1 (Experimental): Single dose A1 of ACT-1014-6470; soft capsule for oral use.
  Interventions: Drug: ACT-1014-6470 (SAD); Drug: Placebo (SAD)
- Part A (SAD): Dose A2 (Experimental): Single dose A2 of ACT-1014-6470; soft capsule for oral use.
  Interventions: Drug: ACT-1014-6470 (SAD); Drug: Placebo (SAD)
- Part A (SAD): Dose A3 (Experimental): Single dose A3 of ACT-1014-6470 under fasted and fed conditions, separated by at least 18 days; soft capsule for oral use.
  Interventions: Drug: ACT-1014-6470 (SAD); Drug: Placebo (SAD)
- Part A (SAD): Dose A4 (Experimental): Single dose A4 of ACT-1014-6470; soft capsule for oral use.
  Interventions: Drug: ACT-1014-6470 (SAD); Drug: Placebo (SAD); Drug: 14C-ACT-1014-6470 microtracer; Drug: 14C-ACT-1014-6470 microtracer placebo
- Part A (SAD): Dose A5 (Experimental): Single dose A5 of ACT-1014-6470; soft capsule for oral use.
  Interventions: Drug: ACT-1014-6470 (SAD); Drug: Placebo (SAD)
- Part A (SAD): Dose A6 (Experimental): Single dose A6 of ACT-1014-6470; soft capsule for oral use.
  Interventions: Drug: ACT-1014-6470 (SAD); Drug: Placebo (SAD)
- Part B (MAD): Dose B1 (Experimental): Multiple doses B1 of ACT-1014-6470; soft capsules for oral use.
  Interventions: Drug: ACT-1014-6470 (MAD); Drug: Placebo (MAD)
- Part B (MAD): Dose B2 (Experimental): Multiple doses B2 of ACT-1014-6470; soft capsules for oral use.
  Interventions: Drug: ACT-1014-6470 (MAD); Drug: Placebo (MAD)
- Part B (MAD): Dose B3 (Experimental): Multiple doses B3 of ACT-1014-6470; soft capsules for oral use.
  Interventions: Drug: ACT-1014-6470 (MAD); Drug: Placebo (MAD)
- Part B (MAD): Dose B4 (Experimental): Multiple doses B4 of ACT-1014-6470; soft capsules for oral use.
  Interventions: Drug: ACT-1014-6470 (MAD); Drug: Placebo (MAD)

INTERVENTIONS:
Drug: ACT-1014-6470 (SAD) — Single dose of ACT-1014-6470; soft capsules for oral use.
  Arms: Part A (SAD): Dose A1; Part A (SAD): Dose A2; Part A (SAD): Dose A3; Part A (SAD): Dose A4; Part A (SAD): Dose A5; Part A (SAD): Dose A6
Drug: ACT-1014-6470 (MAD) — Multiple doses of ACT-1014-6470; soft capsules for oral use.
  Arms: Part B (MAD): Dose B1; Part B (MAD): Dose B2; Part B (MAD): Dose B3; Part B (MAD): Dose B4
Drug: Placebo (SAD) — Single dose of matching placebo; soft capsules for oral use.
  Arms: Part A (SAD): Dose A1; Part A (SAD): Dose A2; Part A (SAD): Dose A3; Part A (SAD): Dose A4; Part A (SAD): Dose A5; Part A (SAD): Dose A6
Drug: Placebo (MAD) — Multiple doses of matching placebo; soft capsules for oral use.
  Arms: Part B (MAD): Dose B1; Part B (MAD): Dose B2; Part B (MAD): Dose B3; Part B (MAD): Dose B4
Drug: 14C-ACT-1014-6470 microtracer — Single dose of 14C-ACT-1014-6470 microtracer; soft capsules for oral use.
  Arms: Part A (SAD): Dose A4
Drug: 14C-ACT-1014-6470 microtracer placebo — Single dose of matching placebo; soft capsules for oral use.
  Arms: Part A (SAD): Dose A4

SUMMARY:
A study to examine the safety, tolerability, and pharmacokinetics of single- and multiple-ascending doses of ACT-1014-6470 in healthy subjects

ELIGIBILITY:
General Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
* Healthy male (Part A and B) and female subjects (Part B) aged between 18 and 55 years (inclusive) at Screening.
* Healthy on the basis of medical history, physical examination, cardiovascular assessments, and clinical laboratory tests.
* Male subjects with a partner who might become pregnant must either be vasectomized or agree to practice adequate contraception from admission to the study site until 3 months after dosing, or the partner must consistently and correctly use a highly effective method of contraception.

Inclusion Criteria for Part B:

* Women of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1. They must consistently and correctly use a highly effective method of contraception with a failure rate of < 1% per year, be sexually inactive, or have a vasectomized partner.
* Women of non-childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1.

General Exclusion Criteria:

* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatment.

Exclusion Criteria for the ADME evaluation (Part A) only:

* Radiation exposure, excluding background radiation but including diagnostic X-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. Occupationally exposed workers, as defined in the relevant Ionising Radiation Regulations, must not participate in the study.
* Participation in any study involving administration of any 14C radiolabeled compound within the 12 months prior to Screening.

Exclusion Criteria for Part B:

- Pregnant or lactating women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
All cohorts: Area under the plasma concentration-time curve (AUC) from zero to infinity (AUC0-inf) | Total duration of assessments: up to 3 weeks.
  Blood samples for determination of PK parameters will be collected at predefined time points from Day 1 to Day 4 of Part A (SAD, Day 1 to Day 8 for ADME cohort A4) and from Day 1 to Day X+3 of Part B (MAD, with Day X = day of last study treatment administration).

OTHER OUTCOMES:
All cohorts: Maximum plasma concentration (Cmax). | Total duration of assessments: up to 3 weeks.
  Blood samples for determination of PK parameters will be collected at predefined time points from Day 1 to Day 4 of Part A (SAD, Day 1 to Day 8 for ADME cohort A4) and from Day 1 to Day X+3 of Part B (MAD, with Day X = day of last study treatment administration)
All cohorts: Time to reach Cmax (tmax). | Total duration of assessments: up to 3 weeks.
  Blood samples for determination of PK parameters will be collected at predefined time points from Day 1 to Day 4 of Part A (SAD, Day 1 to Day 8 for ADME cohort A4) and from Day 1 to Day X+3 of Part B (MAD, with Day X = day of last study treatment administration)
All cohorts: t½. | Total duration of assessments: up to 3 weeks.
  Blood samples for determination of PK parameters will be collected at predefined time points from Day 1 to Day 4 of Part A (SAD, Day 1 to Day 8 for ADME cohort A4) and from Day 1 to Day X+3 of Part B (MAD, with Day X = day of last study treatment administration)
Food effect evaluation only: AUC0-inf under fasted conditions. | Total duration of assessments: up to 3 weeks.
  Blood samples for determination of PK parameters will be collected at predefined time points from Day 1 to Day 4 of Part A (SAD)
Food effect evaluation only: Cmax under fasted conditions. | Total duration of assessments: up to 3 weeks.
  Blood samples for determination of PK parameters will be collected at predefined time points from Day 1 to Day 4 of Part A (SAD)
Food effect evaluation only: tmax under fasted conditions. | Total duration of assessments: up to 3 weeks.
  Blood samples for determination of PK parameters will be collected at predefined time points from Day 1 to Day 4 of Part A (SAD)
Food effect evaluation only: t½ under fasted conditions | Total duration of assessments: up to 3 weeks.
  Blood samples for determination of PK parameters will be collected at predefined time points from Day 1 to Day 4 of Part A (SAD)
Part B (MAD): AUC during a dosing interval (AUCτ) following the first and the last dose. | Total duration of assessments: up to 3 weeks.
  Blood samples for determination of PK parameters will be collected at predefined time points from Day 1 to Day X+3 of Part B (MAD, with Day X = day of last study treatment administration)
Treatment-emergent adverse events (AEs) | Total duration of assessments: up to 3 weeks.
  From start of study treatment administration up to End-of-Study (EOS) or End-of-Period (EOP). - Treatment-emergent serious AEs from the start of the study treatment administration up to EOS or EOP.
Treatment-emergent serious adverse events (SAEs) | Total duration of assessments: up to 3 weeks.
  From start of study treatment administration up to End-of-Study (EOS) or End-of-Period (EOP). - Treatment-emergent serious AEs from the start of the study treatment administration up to EOS or EOP.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No